CLINICAL TRIAL: NCT07206173
Title: Evaluation of the Validity and Reliability of the Londrina Activities of Daily Living Protocol in Patients With Pulmonary Hypertension
Brief Title: Londrina Activities of Daily Living Protocol in Pulmonary Hypertension
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Pinar BASTURK MERC, Principal Investigator, Physiotherapist, PhD, Saglik Bilimleri Universitesi
Other Study IDs: 2459
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Hypertension
Keywords: Londrina Activities of Daily Living Protocol; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Londrina Activites of Daily Living Protocol — The Londrina Activites of Daily Living Protocol is a performance-based test protocol that objectively evaluates ADL. The participant was instructed to perform the tasks at the stations at the same speed they would typically do at home. The protocol consists of five stations with different tasks consisting of arranging objects, walking with weights, organizing objects, organizing clothes and walking.

SUMMARY:
The aim of this observational study is to evaluate the validity and reliability of the Londrina Daily Living Activities Protocol in patients diagnosed with pulmonary hypertension (PH).

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a progressive cardiopulmonary disorder characterized by elevated pulmonary artery pressure, which can lead to right ventricular dysfunction and ultimately heart failure. Right heart catheterization is used to diagnose the disease, and individuals are diagnosed with PH when the mean pulmonary artery pressure is 20 mmHg or higher. The most common and most prominent symptom at diagnosis that prompts referral of PH patients for medical intervention is dyspnea. Dyspnea affects even mild cases of PH, and exertional dyspnea is present in most patients. This significantly impacts patients' functional capacity, quality of life, and overall survival. Even in mild PH, numerous pathological changes contribute significantly to exercise limitation. The multifactorial pathophysiology of exercise limitation in PH involves the circulatory, respiratory, and peripheral muscle systems.

Given the multifaceted nature of pulmonary hypertension and its profound effects on daily functioning, a comprehensive assessment tool is needed to accurately evaluate daily living activities in this patient population. Accurate and reliable assessment of activities of daily living (ADL) is of great importance in the management of pulmonary hypertension, considering the impact of the disease on function. Decreased exercise tolerance in PH, along with reduced quality of life, including physical function and mental health, and decreased physical activity levels, affects every aspect of daily life, placing a significant "disease burden" on the patient.

Quality of life can be assessed primarily using two methods: performance-based tests, which observe the individual's performance while performing standardized activities, and questionnaires, which measure limitations based on the individual's own statements. Performance-based tests offer the advantage of observing the individual's actual performance and identifying potential limitations that may occur during these activities.

The Londrina Activities of Daily Living Protocol is an assessment protocol that aims to evaluate daily living activities and has undergone validity and reliability studies in diseases such as chronic obstructive pulmonary disease, systemic sclerosis, and asthma.

The aim of this study is to evaluate the validity and reliability of the Londrina Activities of Daily Living Protocol in PH.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with pulmonary hypertension (PH)
* Being 18 years of age or older
* Agreeing to participate in the study

Exclusion Criteria:

* Acute decompensated heart failure
* Orthopedic or neurological disorders that prevent the test from being performed
* Patients who have difficulty understanding the instructions given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being diagnosed with pulmonary hypertension (PH)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Londrina Activities of Daily Living Protocol | 15 minutes
  The Londrina ADL protocol will be performed. This protocol consists of a total of 5 stations containing different tasks (arranging objects, walking with weights, organizing objects, organizing clothes and walking). Participants will be asked to perform the tasks at these stations at the speed they would perform them in real life. The duration of the protocol will be recorded in seconds.
  The protocol will be repeated using the same method as the initial evaluation after the patient has rested for at least 30 minutes.
VO2 (ml/kg/min) | 15 minutes
  The Londrina ADL protocol will be performed with a mobile ergospirometer (K5, Cosmed). Oxygen consumption (VO2) obtained during the protocol will be recorded.
  The protocol will be repeated using the same method as the initial evaluation after the patient has rested for at least 30 minutes.

SECONDARY OUTCOMES:
London Chest Activities of Daily Living Scale | 5 minutes
  It is a questionnaire consisting of fifteen items. Each item is given a score ranging from 0 to 5. Higher scores indicate greater limitation in activities of daily living. The total score can reach a maximum of 75
Functional capacity | 6 minutes
  The 6-minute walk test will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The sharing of this information is restricted by the ethics committee and informed consent form.